CLINICAL TRIAL: NCT00884520
Title: An Exploratory, Open Label, Multi-Center, Non-Randomized Study of [F-18]VM4-037
Acronym: VM4-037
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Kirsten Saboe, Clinical Trials Monitor, Clinical Development, Siemens Molecular Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DVM4000
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Lung Cancer; Squamous Cell Carcinoma; Head and Neck Cancer; Hepatic Carcinoma; Renal Cell Carcinoma
Keywords: [F-18]VM4-037; VM4-037; hypoxia; CA-IX; CAIX; carbonic anhydrase IX; hypoxia marker; lung cancer; renal carcinoma; squamous cell carcinoma; hepatic carcinoma; head and neck cancer; advanced stage lung cancer; exploratory
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Squamous Cell; Head and Neck Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Hypoxia | interventions — 3-(4-(2-fluoroethoxy)phenyl)-2-(3-methyl-2-(4-((2-sulfamoylbenzo(d)thiazol-6-yloxy)methyl)-1H-1,2,3-triazol-1-yl)butanamido)propanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VM4-037 (Experimental): Approximately sixteen (16) adult subjects including four (4) healthy volunteers and twelve (12) cancer subjects who have confirmed or highly suspected diagnosis of head & neck, lung, large solitary hepatic and renal cell cancer, as defined by protocol criteria
  Interventions: Drug: [F-18] VM4-037

INTERVENTIONS:
Drug: [F-18] VM4-037 — The individual doses of [F-18]VM4-037 contain a maximum of 20 mCi for normal volunteers and 10 mCi for cancer subjects.
  The single IP dose is administered to the study subject immediately prior to the start of PET imaging.
  Other Names: VM4-037

SUMMARY:
Phase: Exploratory Study

Objectives: To collect drug bio-distribution data, begin collection of baseline and tumor/background imaging data, acquire experience to improve study design and the conduct of future studies

Design: Exploratory, open label, nonrandomized, multi-center study

Duration: Three visits - one screening, one imaging, and one follow-up visit at 24 hours post-dose

Procedures: Informed consent, collection of demographic information and medical history, physical examinations, vital signs, 12-lead ECGs, routine blood tests to assess major organ functions, complete blood counts and clinical chemistries for safety, blood sample for CA-IX assay, pre-dose and post-dose blood samples for metabolite analysis, dosing with [F-18]VM4-037, PET imaging scan, dosimetry estimation (normals), urine collections (normals), tumor immunohistochemistry with CA-IX biomarker, follow up to imaging to collect adverse events

Subjects: Approximately sixteen (16) adult subjects including four (4) healthy volunteers and twelve (12) cancer subjects who have confirmed or highly suspected diagnosis of head & neck, lung, large solitary hepatic and renal cell cancer, as defined by protocol criteria

DETAILED DESCRIPTION:
[F-18]VM4-037 is being developed as a diagnostic radiopharmaceutical for PET imaging.

SMI is seeking to determine if [F-18]VM4-037 might be useful as a PET ligand for the in vivo imaging of CA-IX levels in human tissue.

CA-IX is a very active enzyme which may acidify the extracellular microenvironment of tumor cells in response to hypoxia. Its expression usually promotes tumor growth and invasion, and thus impairs prognosis.

VM4-037 presents no known risks from either in vitro study in cell lines or in vivo study in animals according to in-house preclinical investigations of this compound.

The population to be studied consists of a total of approximately sixteen (16) adult subjects, which includes four normal, healthy volunteers and twelve cancer subjects with a confirmed or highly suspected diagnosis of head and neck cancer, non-small cell lung cancer, large solitary hepatic carcinoma, and renal cell carcinoma as defined by the protocol criteria.

This initial trial will be an Exploratory, Phase 0 study designed to evaluate biodistribution, collect baseline and tumor/background imaging data, and gather preliminary safety data for this investigational product. The study results will be analyzed and considered in the design of future clinical trials.

The primary objectives of this exploratory study are:

* To gain information on the bio-distribution of [F-18]VM4-037, to evaluate the PET images of [F-18]VM4-037 for resolution and signal to background ratio for tumors, and to determine CA-IX expression in tumor tissues by CA-IX antibody with immunohistochemistry
* To collect safety data, and to use this eIND in order to obtain the necessary information to file an IND (Investigational New Drug) application with the FDA (Food and Drug Administration)

The secondary objectives for this exploratory study are:

* To begin collection of baseline imaging and metabolism data
* To gain information to improve study design for the conduct of future trials

The trial is expected to begin subject enrolment in approximately April, 2009 and end subject participation in approximately September, 2009, depending on the rate of enrollment.

The subject is expected to attend three visits, adding up to several hours.

The Investigational Product (IP) being tested in this study is [F-18]VM4-037. The [F-18]VM4-037 will be administered to each qualified subject via a bolus intravenous (IV) injection. For normal volunteers, the dose will not exceed 20 mCi, as the imaging time for dosimetry is a minimum of four hours. For cancer subjects, the dose will be closer to 10 mCi (total imaging time for cancer subjects is about 2 hours).

The procedures for this study include the following:

Obtain Informed Consent, Assign Study Subject Number, Obtain Medical History, Perform Eligibility Blood Labs, Take Pre-Dose Blood Sample for CA-IX Test, Perform Pre-Dose ECG, Monitor and Collect Adverse Events, Collect Concomitant Medications, Perform Pre-Dose Physical Exam, Perform Pre-Dose ECG, Insert IV Line, Take Pre-Dose CBC and Chemistry Blood Labs, Take Pre-Dose Blood Sample for Metabolite Analysis (if applicable), Take Pregnancy Test (if applicable), Take Pre-Dose Vital Signs, Prepare and Administer IP, Perform [F-18]VM4-037 PET Imaging, Take Post-Dose Blood Samples for Metabolite Analysis (if applicable), Take Post-Dose Vital Signs, Perform Post-dose ECGs, Collect Urine Sample and Count for Dosimetry (normal only), Monitor Adverse Events, Collect Concomitant Medications, Perform Physical Exam 24 hr Post-Dose, Take Blood Sample for CBC and Chemistry Labs 24 hr Post-Dose, Perform ECG 24 hr Post-Dose, Take Vital Signs 24 hr Post-Dose, Monitor and Collect Adverse Events, Collect Concomitant Medications, [F-18]FDG PET Imaging, Immunohistochemistry

ELIGIBILITY:
Inclusion Criteria:

Normal Volunteers

* Subject is ≥ 18 years old at the time of investigational product administration, and subject is male or female of any race / ethnicity
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of complying with study procedures
* Subject is capable of communicating with study personnel
* Subject must have renal and hepatic functions and haematological values as defined by laboratory results within defined ranges

Cancer Subjects

* Subject is ≥ 18 years old at the time of the investigational product administration, and subject is a male or female of any race/ethnicity
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of complying with study procedures
* Subject is capable of communicating with study personnel
* Subject must have renal and hepatic functions and haematological values as defined by laboratory results within defined ranges
* Subject must have confirmed or highly suspected non-small cell lung cancer (local or with metastases), squamous cell carcinoma (advanced stages) of the head and neck whose primary origin was from oral cavity, oropharynx, hypopharynx or larynx (local or with metastases), large solitary hepatic carcinoma (primary or metastatic), or renal cell carcinoma (local or with metastases )
* Subject has an adequate size of tumors (≥2 cm) that should be amenable to imaging and biopsy for immunohistochemistry assay using CA-IX and/or hypoxia biomarkers
* Subject did not have any anticancer treatment intervention between [F-18]VM4-037 scan and sampling of biopsied tissue
* Subject is scheduled for a clinical [F-18]FDG PET scan within 14 days either prior to or after the investigational, [F-18]VM4-037 scan (with no anticancer treatment interventions between the two PET scans)
* Subject has a value of ≥ 60% at the time screening according to the Karnofsky Performance Status Scale

Exclusion Criteria:

Normal Volunteers

* Subject is < 18 years old at the time of investigational product administration
* Subject is nursing
* Female subject is pregnant
* Subject is unable to remain still for duration of imaging procedure
* Subject has a significant hepatic or renal disease as defined by previous medical history or abnormal renal and hepatic functions determined by above lab tests in inclusion criteria
* Subject has previously received [F-18]VM4-037 at any time
* Subject has been involved in an investigative, radioactive research procedure within the past 14 days
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality
* Subject has a history of significant prescription or non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives

Cancer Subjects

* Subject is < 18 years old at the time of investigational product administration
* Subject is nursing
* Female subject is pregnant
* Subject is unable to remain still for duration of imaging procedure
* Subject has significant hepatic or renal disease as defined by previous medical history or abnormal renal and hepatic functions determined by above lab tests in inclusion criteria
* Subject has previously received [F-18]VM4-037 at any time
* Subject has been involved in an investigative, radioactive research procedure within the past 14 days
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality
* Subject has a history of significant prescription or non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives
* Subject has had an anticancer treatment intervention between [F-18]VM4-037 scan and biopsied tissue sampling
* Subject has had an anticancer treatment intervention between [F-18]VM4-037 scan and [F-18]FDG scan
* Subject has an inadequate tumor sites or volume (< 2 cm) to allow for PET images and biopsy for immunohistochemistry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety will be the outcome demonstrated in this clinical trial through analyses of adverse events in subjects who receive study drug. | (3) study visits, including the initial screening visit, the imaging visit, and the 24 hour follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yu, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Doss M, Kolb HC, Walsh JC, Mocharla VP, Zhu Z, Haka M, Alpaugh RK, Chen DY, Yu JQ. Biodistribution and radiation dosimetry of the carbonic anhydrase IX imaging agent [(18) F]VM4-037 determined from PET/CT scans in healthy volunteers. Mol Imaging Biol. 2014 Oct;16(5):739-46. doi: 10.1007/s11307-014-0730-7. PMID 24696183